CLINICAL TRIAL: NCT01963351
Title: Open-label Study of Bevacizumab (AVASTIN®) in Combination With Platinum-containing Chemotherapy as First-line Treatment of Patients With Advanced or Recurrent Non-squamous Non-small Cell Lung Cancer
Brief Title: Bevacizumab in Combination With Chemotherapy in Patients With Advanced or Recurrent Non-squamous NSCLC
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Kostas N Syrigos, Professor in Medical Oncology, University of Athens
Other Study IDs: ML27816
Record Dates: First submitted 2013-09-19; First posted 2013-10-16 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Non-small Cell Lung Cancer; Unresectable Malignant Neoplasm
Keywords: NSCLC; Non-squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Locally advanced and metastatic nsclc: non squamous

SUMMARY:
This observational trial is designed to assess the safety profile and tolerability of bevacizumab when combined with chemotherapy as first-line treatment of advanced or recurrent non-squamous NSCLC.

DETAILED DESCRIPTION:
It is an observational study for the safety and tolerability of the combination of bevacizumab with chemotherapy in locally advanced or metastatic and recurrent non-squamous non-small cell lung cancer. We try to evaluate the safety of bevacizumab in real life population with lung cancer. For patients with performance status 0-1 platinum based chemotherapy was recommended and acceptable doses of bevacizumab was either 7.5 or 15 mg/kgr. Safety profile was evaluated with Common Toxicity criteria v 3.0. Especially for bevacizumab we evaluate specific situations as thrombotic or hemorrhagic events, hypertension, albuminuria, and gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent 2. Age ≥18 years 3. Able to comply with the protocol 4. Histologically or cytologically documented, locally advanced, metastatic (Stage IV) or recurrent non-squamous NSCLC 5.ECOG PS: 0-2 6. Life expectancy ≥12 weeks 7. Adequate haematological function:
* Absolute neutrophil count (ANC) ≥1.5 x 109/L AND
* Platelet count ≥100 x 109/L AND
* Haemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level) 8. Adequate liver function:
* Total bilirubin <1.5 x upper limit of normal (ULN) AND
* Asparagine aminotransferase (AST), alanine aminotransferase (ALT) <2.5 x ULN in patients without liver metastases; <5 x ULN in patients with liver metastases 9. Adequate renal function: calculated creatinine clearance ≥50 mL/min AND
* Urine dipstick for proteinuria <2+. 10. INR ≤1.5 and partial prothrombin time (PTT or aPTT) ≤1.5 x ULN within 7 days prior to enrolment 11. If female, should not be pregnant or breast-feeding. Women with an intact uterus (unless amenorrhoeic for the last 24 months) must have a negative serum pregnancy test within 28 days prior to enrolment into the study

Exclusion Criteria:

1. Mixed, predominant squamous component
2. History of haemoptysis, in the 3 months prior to enrolment
3. Evidence of tumour invading major blood vessels
4. Evidence of CNS metastases, even if previously treated. If suspected, the patient should be scanned within 28 days prior to enrolment to rule out CNS metastases
5. Neoadjuvant/adjuvant chemotherapy within 6 months prior to enrolment
6. Radical radiotherapy with curative intent within 28 days prior to enrolment. Palliative radiotherapy f is allowed
7. Major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrolment
8. Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion
9. Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (> 325mg/day)
10. Current or recent use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes. Prophylactic use of anticoagulants is allowed
11. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
12. Uncontrolled hypertension
13. Clinically significant (i.e. active) cardiovascular disease
14. Non-healing wound, active peptic ulcer or bone fracture
15. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment
16. Women with an intact uterus (unless amenorrhoeic for the last 24 months) not using effective, means of contraception Men who do not agree to use effective contraception during the study

18. Known hypersensitivity to bevacizumab or any of its excipients, and any of the chemotherapies 19. Evidence of ongoing or active infection, any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications 20. Patients diagnosed with a tracheo-esophageal fistula 21. Prior chemotherapy or treatment with another systemic anti-cancer agent 22. Malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, DCIS treated surgically with curative intent 23. History of thrombotic disorders within the last 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically documented advanced metastatic (patients who are not candidates for radiotherapy, i.e. supraclavicular lymph node metastases or Stage IIIb with malignant pleural or pericardial effusion or Stage IV) or recurrent non-squamous non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events during 24 months of follow-up | 24 months

SECONDARY OUTCOMES:
Overall survival | 24 months

OTHER OUTCOMES:
Progression free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kostas N Syrigos, Professor, Study Chair — Oncology Unit University of Athens, Sotiria Hosp, 152 Mesogion Av
Locations (1):
- Oncology Unit Sotiria Hospital of Chest Diseases, Athens, Greece